CLINICAL TRIAL: NCT06233916
Title: Mass Balance Study of [14C] D-1553 in Chinese Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D1553-108
Record Dates: First submitted 2023-11-27; First posted 2024-01-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Mass Balance Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C] D-1553 group (Other): Single arm study
  Interventions: Drug: [14C] D-1553

INTERVENTIONS:
Drug: [14C] D-1553 — [14C] D-1553 (approximately 400 mg/80 μCi)

SUMMARY:
* To quantitatively analyze the total radioactivity (TRA) in excrement after a single oral dose of [14C] D-1553 in healthy subjects, and obtain radioactivity recovery and primary excretion pathways in humans;
* To obtain radioactive metabolite profiles of human plasma, urine and feces , identify major metabolites of D-1553 and determine the major metabolic pathways and elimination pathways;
* To quantitatively analyze the TRA in whole blood and plasma and obtain PK parameters of plasma TRA and investigate whole blood/plasma ratio for TRA.

DETAILED DESCRIPTION:
Primary Objectives:

* To quantitatively analyze the total radioactivity (TRA) in excrement after a single oral dose of [14C] D-1553 in healthy subjects, and obtain radioactivity recovery and primary excretion pathways in humans;
* To obtain radioactive metabolite profiles of human plasma, urine and feces after a single oral dose of [14C] D-1553 in healthy subjects, identify major metabolites of D-1553 and determine the major metabolic pathways and elimination pathways;
* To quantitatively analyze the TRA in whole blood and plasma after a single oral dose of [14C] D-1553 in subjects, and obtain PK parameters of plasma TRA and investigate whole blood/plasma ratio for TRA.

Secondary Objectives:

* To observe the safety of a single oral dose of [14C] D-1553 in healthy subjects;
* To quantitatively analyze the concentration of D-1553 and its metabolites (if applicable) in plasma using the validated LC-MS (liquid chromatography-mass spectrometry)/MS method and obtain the pharmacokinetic (PK) parameters of D-1553 and its metabolites (if applicable) in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who volunteer to participate in this clinical trial, understand the study procedures and sign the Informed Consent Form (ICF) in writing.
* Healthy Chinese adult male subjects aged 19-55 years (inclusive) at the time of signing the ICF.
* Body weight ≥ 50.0 kg, 19 kg/m2 ≤ body mass index (BMI) ≤ 26.0 kg/m2, and BMI = body weight (kg)/body height2 (m2) at screening.
* Subjects with normal test results or with abnormal but not clinically significant results as judged by the clinician for vital signs, physical examination, 12-lead ECG, chest radiograph (PA view), abdominal color Doppler ultrasound (liver, gallbladder, pancreas, spleen, and kidneys), ophthalmological examination, and laboratory tests (including hematology, blood chemistry, coagulation function, urinalysis, thyroid function, screening for infectious diseases, stool routine test + occult blood) during screening.
* Subjects who agree to abstain, are surgically sterilized, or agree to use an effective contraceptive method from the time of signing the ICF and for the duration of study participation to 180 days after administration of the study drug.

Exclusion Criteria:

* Subjects with any medical history of disorders of the central nervous system, cardiovascular system, blood and lymphatic system, immune system, urinary system, digestive system, respiratory system, and metabolic and skeletal system, etc., other acute or chronic diseases or mental diseases, which are abnormal and clinically significant at the discretion of the investigator.
* Subjects who are positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody, treponema pallidum antibody (TPA), or HIV antigen/antibody combination test (preliminary screening).
* Subjects who have smoked more than 5 cigarettes or 1 pipe per day (or equivalent of nicotine products) on average within 3 months prior to screening, or who are unable to stop using any tobacco products during the trial.
* Subjects with hemorrhoids with hematochezia or perianal disease with regular/ongoing hematochezia, or with severe nausea, vomiting, constipation or diarrhea within one week prior to screening; or with positive test results for fecal occult blood.
* Subjects with a history of blood or needle phobia.
* Subjects who have undergone a major surgery that affects the absorption or metabolism of the study drug within 6 months prior to the first dose.
* Subjects who have participated in clinical trials of other study drugs within 3 months before the first dose; if the half-life of that other investigational drug is long, the time period is limited to 5 half-lives of the drug.
* Subjects unwilling or unable to follow the life restrictions described in the study protocol (such as dietary restrictions, activity and contraceptive requirements, etc.).
* Subjects who have lost blood or donated blood, or received blood transfusions or used blood products within 1 month before administration.
* Subjects who are exposed to radioactive work conditions for a long time, or have significant radiation exposure (≥ 2 chest/abdominal CTs, or ≥ 3 other types of X-ray examinations) within 1 year before the first dose, or have participated in a radiopharmaceutical labeled trial.
* Subjects who are unsuitable for the study participation for other reasons at the discretion of the investigator.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Chinese adult male subjects aged 19-55 years (inclusive) at the time of signing the ICF.
Enrollment: 8 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
The radioactivity will be determined by a liquid scintillation counter. Analyze the total recovery (that is the ratio of the radioactivity in excrement samples to the radioactivity of the drug that administered ) in excrement | 2 weeks
  Recovery and cumulative recovery of total radioactive substance in excrement (urine and feces)
Percentage of unchanged drug and its metabolites in plasma, urine and feces to the administered dose | 2 weeks
  Exposure in plasma; percentage of unchanged drug and its metabolites in urine and feces to the administered dose; identification of major metabolites in plasma, urine and feces
whole blood/plasma ratio for TRA (total radioactivity) concentration at different time points | 2 weeks
  whole blood/plasma ratio for TRA concentration at different time points
Tmax (time to maximum observed concentration) parameters of TRA; | baseline to 2 weeks
  Tmax parameters of TRA in plasma
t1/2 (terminal elimination half-life) parameters of TRA; | baseline to 2 weeks
  t1/2 parameters of TRA in plasma
Cmax (maximum concentration) parameters of TRA; | baseline to 2 weeks
  Cmax parameters of TRA in plasma
MRT (mean residence time) parameters of TRA; | baseline to 2 weeks
  MRT parameters of TRA in plasma
AUC (area under curve) parameters of TRA; | baseline to 2 weeks
  AUC parameters of TRA in plasma

SECONDARY OUTCOMES:
Incidence and severity of AEs based on NCI CTCAE V5.0 | baseline to 3 weeks
  Incidence and severity of adverse events (AEs) graded based on NCI CTCAE V5.0
Incidence and severity of SAEs based on NCI CTCAE V5.0 | baseline to 3 weeks
  Incidence and severity of serious adverse events (SAEs) graded based on NCI CTCAE V5.0
Tmax parameters of D-1553 and its metabolites | baseline to 2 weeks
  Tmax parameters of D-1553 and its metabolites (if applicable) in plasma
Cmax parameters of D-1553 and its metabolites | baseline to 2 weeks
  Cmax parameters of D-1553 and its metabolites (if applicable) in plasma
AUC0-t parameters of D-1553 and its metabolites | baseline to 2 weeks
  AUC0-t parameters of D-1553 and its metabolites (if applicable) in plasma
T1/2 parameters of D-1553 and its metabolites | baseline to 2 weeks
  T1/2 parameters of D-1553 and its metabolites (if applicable) in plasma
MRT parameters of D-1553 and its metabolites | baseline to 2 weeks
  MRT parameters of D-1553 and its metabolites (if applicable) in plasma
CL/F (apparent clearance) parameters of D-1553 and its metabolites | baseline to 2 weeks
  CL/F parameters of D-1553 and its metabolites (if applicable) in plasma
Vz/F (apparent volume of distribution) parameters of D-1553 and its metabolites | baseline to 2 weeks
  Vz/F parameters of D-1553 and its metabolites (if applicable) in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- beijing Gobroad Boren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No